CLINICAL TRIAL: NCT07199907
Title: Hippocampal and Frontoparietal Mechanisms of Knowledge Acquisition and Inference
Brief Title: Hippocampal and Frontoparietal Development and Inference
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Nicole Varga (Unknown)
Responsible Party: Principal Investigator, Alison Preston, Professor, University of Texas at Austin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012090055; 5R01MH100121 (NIH)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Hippocampus; Medial Prefrontal Cortex; Parietal Cortex; Memory; Reasoning; Inference; Adolescence; Brain Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescents (Experimental): Participants completed a predictable (associative inference; Session 1) and noisy (probabilistic inference; Session 2) learning task during fMRI scanning. Participants completed these tasks three times, once every 18 months.
  Interventions: Behavioral: Associative Inference; Behavioral: Probabilistic Inference
- Adults (Experimental): Participants completed a predictable (associative inference; Session 1) and noisy (probabilistic inference; Session 2) learning task during fMRI scanning. Participants completed these tasks a single time, serving as a control comparison to our adolescent arm.
  Interventions: Behavioral: Associative Inference; Behavioral: Probabilistic Inference

INTERVENTIONS:
Behavioral: Associative Inference — Objects, faces, and scenes will be arranged into 12 ABC triads presented as overlapping AB and BC pairs. AB pairs will comprise objects; BC pairs will consist of the same B object paired with a face or scene (C). Twelve non-overlapping (NO) pairs will serve as controls. Participants will study overlapping (AB, BC) and NO pairs (4s) across two 5-minute fMRI runs. Each pair will be presented three times within a run. Following learning, participants will complete a self-paced 3-alternative forced choice (AFC) inference task during which they will select the C item that shares a common relationship with an A cue. Foils for inference trials will be C items from other ABC triads, of the same face/scene subcategory. Participants will then complete a final, self-paced 3-AFC memory test of premise associations (AB, BC) and NO pairs. To quantify memory retrieval and how overlapping events are organized, before and after learning, participants will view the A and C items during fMRI scanning.
Behavioral: Probabilistic Inference — Participants will visit a virtual "zoo," which is divided into three zones, each containing the same five monsters, but with different likelihoods of occurrence. Participants learn the underlying likelihood distributions by virtually navigating each zone. On each trial, two monsters appear; participants select the monster that they predict will next appear (6s). After making their choice, the correct monster appears and feedback is provided (2s). Participants tour each zone four times across 9 runs. Following learning, participants are tested on probabilistic inference. Here, participants see a series of monster "photographs" and are asked to infer in which zone they were taken. On each trial, a sequence of individual monster images (3.5s each) will then appear (1-6 monsters) prior to a decision screen, in which participants choose which of the two zones most likely produced the "photos" (4s) and are given feedback (1.5s). Participants will perform nine fMRI runs of the inference task.

SUMMARY:
The goal of this clinical trial is to test if an intervention used to manipulate memory and inference can improve our understanding of how brain development supports these abilities in healthy adolescent and adult volunteers. The main questions it aims to answer are: (1) Do hippocampus and ventromedial prefrontal cortex shift from forming simple memories for singular experiences to more complex memories that link numerous experiences together?; (2) Does an improved ability to retrieve prior memories in parietal cortex during new learning have consequences for how those memories are organized at different ages?; and (3) Does the emerging memory control supported by ventromedial prefrontal cortex development facilitate the formation of optimally-organized memory representations? Adolescent participants (13-18 years) will perform two experimental tasks during functional magnetic resonance imaging (fMRI) scanning at three timepoints (T1-T3), spaced 1.5 years apart. Researchers will compare behavioral and neuroimaging data to a separate group of adults (19-25 years) who will perform the task at a single timepoint (T1). The tasks and comparison groups will allow us to isolate the neural processes that support memory and inference behavior, and how these processes change with age.

DETAILED DESCRIPTION:
Hippocampus (HPC) structure and its connectivity with frontoparietal regions continue to develop through adolescence, a developmental period associated with substantial gains in memory and reasoning. While such structural changes are well documented, we know less about the functions that HPC and frontoparietal development confer, fundamentally limiting our understanding of the mechanisms through which individuals learn and reason about the world at different ages. From very early in life, children can learn simple associations that they directly experience. However, with age, our memories become more complex, reflecting not only directly observed information, but also knowledge derived across multiple episodes. Such derived knowledge might represent commonalities among experiences while simultaneously exaggerating important differences between them, thus forming hierarchical knowledge structures that can support inference decisions about event relationships, while also preserving detailed memory for when and where those relationships vary by context. The overarching goal of this proposal is to test the hypothesis that representational capacity within HPC and frontoparietal cortex undergoes qualitative changes during adolescence. We will use a serial cohort design to collect data from adolescents (13-18 years) at three timepoints, each 1.5 years apart, as well as data from adults (19-25 years) at a single timepoint. This design will allow us to test longitudinal predictions about how changes in neural representation within individual adolescents, over time, predict corresponding changes in memory and inference behaviors, as well as cross-sectional predictions about how HPC and frontoparietal cortex representation differs between adolescents and adults. We will use high-resolution functional magnetic resonance imaging (fMRI), representational fMRI analyses, and computational modeling, to test three Aims. Aim 1 will test the prediction that HPC and ventromedial prefrontal (vmPFC) representations will transition from coding simple, individual associations to extracting hierarchical knowledge about the relationships among experiences. Aim 2 will test the prediction that lateral parietal cortex (LPC)-mediated memory reactivation during new learning and inference will have different consequences for HPC-vmPFC representation and inference behavior at distinct points in adolescence. Aim 3 will test the prediction that emerging vmPFC control will influence what memories are available in LPC during learning and inference, as well as directly mediate the impact reactivated memories have on the trajectory of HPC representation during adolescence. The results from this project will provide a key test of fundamental theories of cognitive development and substantially advance our knowledge of the representational capacities of the HPC-frontoparietal memory system in typically developing adolescents. In doing so, the findings may have important implications for our eventual understanding of how the onset of mental health disorders (e.g., affective disorders and schizophrenia) during adolescence impact neural representation as well as memory and reasoning ability.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Have normal or corrected to normal vision
* Have normal hearing
* Do not have contraindications for MRI
* Have no history of neurological or psychiatric disorders at initial intake
* Are of normal intelligence
* Native or fluent English speaker

Exclusion Criteria:

* A major medical illness or a neurological disorder, or neurological abnormality including significant head trauma (loss of consciousness > 5 min).
* Meeting criteria for any psychiatric disorder or any prior psychiatric hospitalizations
* Intelligence scores more than 1 standard deviation below the mean on the WASI-II
* History of special education placement
* Non-native English speaker
* Prior use of psychotropic medication, except antidepressants, for longer than 1 month
* History of moderate to severe cannabis use disorder, via self-report
* MRI exclusions: Claustrophobia; tattoos above the shoulders; permanent eyeliner; permanent retainer or spacer; artificial eyebrows; cardiac pacemaker; metal fragments in eye, skin, or body, including shrapnel; heart valve replacement; brain clips; venous umbrella; being a sheet-metal worker or welder; lifetime history of aneurysm surgery; intracranial bypass, renal, or aortic clips; prosthetic devices such as middle ear, eye, joint, or penile implants; joint replacements; non-removable hearing aid, neurostimulator, or insulin pump; shunts/stents; metal mesh/coil implants; metal plate/pin/screws/wires; or any other metal implants; or suspected pregnancy.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Changes in blood oxygen-level dependent (BOLD) signal over time | 36 months
  Within the adolescent group, changes in BOLD signal during task performance, as measured by functional magnetic resonance imaging (fMRI), will be assessed across three separate timepoints.
Differences in blood oxygen-level dependent (BOLD) signal between age groups | 1 month
  Differences in BOLD signal during task performance, as measured by functional magnetic resonance imaging (fMRI), will be compared between the adolescent and adult groups at timepoint 1.

SECONDARY OUTCOMES:
Changes in task behavior over time | 36 months
  Within the adolescent group, changes in task performance, as measured by the two behavioral interventions, will be assessed across three separate timepoints.
Differences in task behavior between age groups | 1 month
  Differences in task performance, as measured by the two behavioral interventions, will be compared between the adolescent and adult groups at timepoint 1.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The present research will generate magnetic resonance imaging (MRI) data and associated electronic records of task behavior, standardized assessments, and magnetic resonance images, along with statistical maps of brain regions involved in task performance. Data and analysis code will be shared on public repositories (e.g., OSF, NDA). Data will be formatted in the standard brain imaging data structure (BIDS) format, which includes comprehensive metadata and is compatible with many analysis packages, promoting reuse of data for future projects. Raw neuroimaging data will also be shared on NDA. Results and conclusions will also be shared via peer-reviewed publications and presentations at scientific meetings such as the annual meetings of the Society for Neuroscience, the Cognitive Neuroscience Society, and Flux: The Society for Developmental Cognitive Neuroscience.